CLINICAL TRIAL: NCT05916274
Title: Pro-inflammatory Role of Extracellular DNA in Inflammatory Bowel Disease in Children: Study of the cGAS-STING Pathway
Brief Title: Exploration of the Activity of DNA Located Outside of Cellular Nucleus to Amplify Inflammation in Inflammatory Bowel Disease in Children Through Biological Pathway Cyclic GMP-AMP Synthase (cGAS) - Stimulator of Interferon Genes (STING)
Acronym: ROXANE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHRO-2023-01
Record Dates: First submitted 2023-05-05; First posted 2023-06-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: Inflammatory Bowel disease; Crohn disease; Ulcerative colitis; cell-free DNA; cGAS; STING; Child; intestinal inflammation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Bites and Stings | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with samples (Other): Blood and fecal samples, and colonic biopsies will be analysed and compared between 3 groups of participants :1/ Active IBD; 2/Inactive IBD; 3/Controls "non-IBD".
  Interventions: Biological: Blood and fecal samples; Procedure: Coolonic biopsies

INTERVENTIONS:
Biological: Blood and fecal samples — Blood and fecal samples will be performed
Procedure: Coolonic biopsies — colonic biopsies will be analysed

SUMMARY:
Frequency of Inflammatory Bowel Diseases in children (IBD)-Crohn's disease (CD), Ulcerative colitis (UC) is constantly increasing. Pediatric-onset IBD represent a different nosological entity (from adult IBD) because of their major inflammatory activity, their significant anatomical extent and their stenotic and/or fistulizing character sometimes from diagnosis. Intestinal lesions are due to dysregulation of the intestinal immune system but the cause is unknown. The investigators hypothesize that extranuclear DNA participates in the amplification of the inflammatory response at the intestinal and blood levels during pediatric IBD through the cGAS-STING pathway. The investigators will analyse blood and fecal samples, and colonic biopsies issued from ill children and control participants on age of 6 to 17 years. The investigators think that this study will provide a better understanding of the mechanisms involved in pediatric IBD, assess the place of the cGAS-STING pathway, identify potential biomarkers of pediatric IBD and new potential therapeutic targets based in particular on the inhibition of the cGAS-STING pathway.

DETAILED DESCRIPTION:
Inflammatory Bowel Diseases in children (IBD)-Crohn's disease (CD), ulcerative colitis (UC) are severe pathology that can affect the entire digestive tract. Their annual incidence is however constantly increasing.

IBD are complex multifactorial pathologies whose cause is still unknown today. IBD occurs on a predisposing genetic background in the presence of exogenous factors and alteration of the intestinal microbiota. Intestinal lesions are due to dysregulation of the intestinal immune system with increased secretion of pro-inflammatory cytokines at the expense of anti-inflammatory cytokines.

Pediatric-onset IBD represent a different nosological entity (from adult IBD) because of their major inflammatory activity, their significant anatomical extent and their stenotic and/or fistulizing character sometimes from diagnosis. Their impact is not only individual (growth retardation, puberty delay, psychological disorders) but also family/parental, school and social. These particularities justify that biomedical research focuses on it in a more specific way.

Extracellular and extranuclear DNA (enDNA) play a major role in innate immunity by stimulating pro-inflammatory responses and activating type I interferon production. The pro-inflammatory action of enDNA is mediated by enzyme cGAS, protein STING, toll-like receptor 9 (TLR9), and the inflammasome complex NLRP3.

The investigators hypothesize that enDNA participates in the amplification of the inflammatory response at the intestinal and blood levels during pediatric IBD through the cGAS-STING pathway. They also hypothesize that there are links between the cGAS-STING pathway and other pathways involved in pediatric IBD such as NOD2 and Autophagy. The investigators will analyse blood and fecal samples, and colonic biopsies issued from ill children and controls on age of 6 to 17 years. The investigators think that this study will provide a better understanding of the mechanisms involved in pediatric IBD, assess the place of the cGAS-STING pathway, identify potential biomarkers of pediatric IBD and new potential therapeutic targets based in particular on the inhibition of the cGAS-STING pathway.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged from 6 years inclusive to 17 years inclusive
* Boys and girls
* Presenting an IBD or suspicion of IBD
* Requiring a colonoscopy for diagnosis or follow-up or other reason (abdominal pain, diarrhoea, rectal bleeding, weight loss) not confirming the diagnosis of Crohn's disease or Ulcerative Colitis
* Active IBD if:

  * CD: PCDAI score >5 and CRP>20mg/L and faecal calprotectin> 400 µg/g
  * UC: PUCAI score>10 and faecal calprotectin>250 µg/g
* IBD in remission if:

  * CD: PCDAI score<5 and CRP<20mg/L and faecal calprotectin<400 µg/g
  * UC: PUCAI score <10 and faecal calprotectin < 250 µg/g
* Patients and their parents who gave their consent to participate in the study

Exclusion Criteria:

* Refusal of the participant and/or one of his two parents
* Body weight less than or equal to 20 kg
* Blood hemoglobin level less than or equal to 9 g/dl
* Refusal or contraindication to general anesthesia
* Co-existing severe chronic pathology and/or treatment that could interfere with the results of the study; example: trisomy 21, treatment with growth hormone etc.
* Protected person (under guardianship or curatorship)
* Person under legal protection
* Person not affiliated to a social security scheme
* Pregnant or breastfeeding woman

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Amount of mRNA specific for colonic cGAS | Baseline
  the comparison, between the 3 groups of patients, of the quantity of specific mRNA of colonic cGAS expressed as the number of "reads" during RNA sequencing (RNAseq), by a Mann-Whitney U test. It is planned from the outset to compare the groups 2 by 2, regardless of the result of an overall test such as a Kruskal-Wallis test.

SECONDARY OUTCOMES:
quantitative difference of amount of circulating mtDNA | Baseline
  to find quantitative differences between the 3 groups concerning the circulating mtDNA, the circulating total DNA, by the qPCR technique: by specific primer sequences to identify the origin of the DNA (mitochondrial or nuclear). Results will be expressed by the -2∆∆Ct method ("fold increase") compared to the control.
Cytokine response | Baseline
  to find quantitative differences between the 3 groups concerning the cytokine response by Luminex®: in pg/ml or in ng/ml depending on the cytokines
inflammatory / dysimmune response of cytokines | Baseline
  to find quantitative differences between the 3 groups concerning the inflammatory / dysimmune response of cytokines, components of the cGAS-STING pathways autophagy, NOD2, intestinal mucins, integrins, cadherins by RNAseq type transcriptomic analysis in Transcript Per Million (TPM).
  This outcome wil be mesured at the blood level abd the colonic level.
Difference of DNA methylation by Methyl-Seq between the 3 groups | Baseline
  to find quantitative differences between the 3 groups concerning the study of DNA methylation by Methyl-Seq. Results expessed in pourcentage of methylation. This outcome will be mesured at the bllod level and the colonic level.
Activation (phosphorylation) of the components of the cGAS-STING pathway | Baseline
  Activation (phosphorylation) of the components of the cGAS-STING pathway (proteins cGAS, p-CGAS, STING,p-STING,TBK1, p-TBK1,IRF-3, p-IRF-3) by Western-Blot
plasma DNase activity | baseline
  plasma DNase activity in Kunitz unitz
differences in microbial distribution | Baseline
  search for quantitative differences in microbial distribution between the 3 groups by pyrosequencing RNA 16s of the microbiota at the fecal level
quantity (number of "reads") of colonic STING-specific mRNA | Baseline
  quantitative differences between the 3 groups concerning the quantity (number of "reads") of colonic STING-specific mRNA at the colonic level
extracellular DNA by qPCR | Baseline
  We will use specific primer sequences to identify the origin of the DNA (mitochondrial or nuclear). Results will be expressed by the -2∆∆Ct method ("fold increase") compared to the control. This outcome will be mesured at the colonic level.
Amount of STING in the cytoplasm | Baseline
  cytoplasmic presence of STING by histology, immunohistochemical staining and optical microscopy analysis. Results will be qualitative (present/absent; localization) and quantitative based on optical density (pourcentage of positive cells)
Amount of cGAS in the cytoplasm | Baseline
  cytoplasmic presence of cGAS by histology, immunohistochemical staining and optical microscopy analysis. Results will be qualitative (present/absent; localization) and quantitative based on optical density (pourcentage of positive cells)
Amount of nuclear DNA in teh cytoplasm | Baseline
  cytoplasmic presence of nuclear DNA by histology, immunohistochemical staining and optical microscopy analysis. Results will be qualitative (present/absent; localization) and quantitative based on optical density (pourcentage of positive cells)
Amount of mitochondrial DNA in the cytoplasm | Baseline
  cytoplasmic presence of mitochondrial DNA by histology, immunohistochemical staining and optical microscopy analysis. Results will be qualitative (present/absent; localization) and quantitative based on optical density (pourcentage of positive cells)
Amount of colonic DNase activity | Baseline
  Measurement of colonic DNase activity in Kunitz unitz

CONTACTS AND LOCATIONS:
Overall Officials: Georges DIMITROV, MD, Principal Investigator — CHU Orleans
Locations (1):
- CHU Orléans, Orléans, France

REFERENCES:
- [Background] Ahn J, Son S, Oliveira SC, Barber GN. STING-Dependent Signaling Underlies IL-10 Controlled Inflammatory Colitis. Cell Rep. 2017 Dec 26;21(13):3873-3884. doi: 10.1016/j.celrep.2017.11.101. PMID 29281834
- [Background] Canesso MCC, Lemos L, Neves TC, Marim FM, Castro TBR, Veloso ES, Queiroz CP, Ahn J, Santiago HC, Martins FS, Alves-Silva J, Ferreira E, Cara DC, Vieira AT, Barber GN, Oliveira SC, Faria AMC. The cytosolic sensor STING is required for intestinal homeostasis and control of inflammation. Mucosal Immunol. 2018 May;11(3):820-834. doi: 10.1038/mi.2017.88. Epub 2017 Dec 20. PMID 29346345
- [Background] Martin GR, Blomquist CM, Henare KL, Jirik FR. Stimulator of interferon genes (STING) activation exacerbates experimental colitis in mice. Sci Rep. 2019 Oct 3;9(1):14281. doi: 10.1038/s41598-019-50656-5. PMID 31582793
- [Background] Boyapati RK, Dorward DA, Tamborska A, Kalla R, Ventham NT, Doherty MK, Whitfield PD, Gray M, Loane J, Rossi AG, Satsangi J, Ho GT. Mitochondrial DNA Is a Pro-Inflammatory Damage-Associated Molecular Pattern Released During Active IBD. Inflamm Bowel Dis. 2018 Sep 15;24(10):2113-2122. doi: 10.1093/ibd/izy095. PMID 29718255
- [Background] Vrablicova Z, Tomova K, Tothova L, Babickova J, Gromova B, Konecna B, Liptak R, Hlavaty T, Gardlik R. Nuclear and Mitochondrial Circulating Cell-Free DNA Is Increased in Patients With Inflammatory Bowel Disease in Clinical Remission. Front Med (Lausanne). 2020 Dec 14;7:593316. doi: 10.3389/fmed.2020.593316. eCollection 2020. PMID 33381513
- [Background] Khan S, Mentrup HL, Novak EA, Siow VS, Wang Q, Crawford EC, Schneider C, Comerford TE 4th, Firek B, Rogers MB, Loughran P, Morowitz MJ, Mollen KP. Cyclic GMP-AMP synthase contributes to epithelial homeostasis in intestinal inflammation via Beclin-1-mediated autophagy. FASEB J. 2022 May;36(5):e22282. doi: 10.1096/fj.202200138R. PMID 35344224
- [Background] Zhao F, Zheng T, Gong W, Wu J, Xie H, Li W, Zhang R, Liu P, Liu J, Wu X, Zhao Y, Ren J. Extracellular vesicles package dsDNA to aggravate Crohn's disease by activating the STING pathway. Cell Death Dis. 2021 Aug 27;12(9):815. doi: 10.1038/s41419-021-04101-z. PMID 34453041
- [Background] Chen C, Zhang Y, Tao M, Zhao X, Feng Q, Fei X, Fu Y. Atrial Natriuretic Peptide Attenuates Colitis via Inhibition of the cGAS-STING Pathway in Colonic Epithelial Cells. Int J Biol Sci. 2022 Feb 7;18(4):1737-1754. doi: 10.7150/ijbs.67356. eCollection 2022. PMID 35280696